CLINICAL TRIAL: NCT04845789
Title: Case Manager Approach in Dementia Care From a Caregiver Perspective: A Grounded Theory Study
Brief Title: Case Manager Approach in Dementia Care From a Caregiver Perspective
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Jockey Club Centre for Positive Ageing (Other)
Responsible Party: Principal Investigator, Lui Kam Yan, Principal investigator, Chinese University of Hong Kong
Other Study IDs: CaseManagerDementiaGT
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Family caregivers: Family caregivers who were main caregiver to the person with dementia and who spent at least 10 hours a week providing care to the person with dementia.
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Non-interventional. Interview would be conducted for data collection.

SUMMARY:
This is a qualitative study to explore opinions of family caregivers of community-dwelling people with dementia on case manager approach in dementia care. Semi-structured interviews will be used for data collection. Purposive sampling was used to recruit caregivers from Jockey Club Centre for Positive Ageing. Grounded Theory would be used for data analysis.

DETAILED DESCRIPTION:
This was a qualitative study using semi-structured interviews with caregivers of community-dwelling people with dementia. Purposive sampling was used to recruit caregivers from Jockey Club Centre for Positive Ageing.

Study protocol would be explained by principal investigator (PI) to case managers in JCCPA, including aim and objectives of the study, inclusion criteria, exclusion criteria and interview questions.

Due to privacy issues, case managers in JCCPA would screen family caregivers and ask for consent to participate in the study. Contact method of caregivers would be provided to PI by JCCPA case managers upon caregivers' consent. PI would then approach caregivers to arrange online meetings and send the online consent form to them for their consideration and reference. Risks and benefits of the study and the right to withdraw from the study at any time would be explained to participants before consent form was signed by participants digitally.

Demographic data such as age, gender, education level, years of caregiving to PWD and time spent on caregiving would be collected using Google form.

All interviews were conducted through video-conferencing individually. Each interview took 30 to 45 minutes. The interviews were started with an close-ended question, such as "Do you know the special approach that JCCPA has adopted?" and "Did the staff tell you about it at admission?", followed up by open-ended questions such as "What do you know about case management?" and "Can you tell me how your caregiving experience was with case manager support?". Subsequent probing questions aimed at clarification and gaining more insight on their experience, was guided by the participant's responses.

Demographic data such as age, gender, education level, years of caregiving to PWD and time spent on caregiving would be collected using Google form.

All interviews were conducted through video-conferencing individually. Each interview took 30 to 45 minutes. The interviews were started with an close-ended question, such as "Do you know the special approach that JCCPA has adopted?" and "Did the staff tell you about it at admission?", followed up by open-ended questions such as "What do you know about case management?" and "Can you tell me how your caregiving experience was with case manager support?". Subsequent probing questions aimed at clarification and gaining more insight on their experience, was guided by the participant's responses. Video-conferencing software such as Zoom, Google Meet, or facetime would be used for online interview. Interview would be conducted in JCCPA to ensure privacy of the participants.

All interviews were audio recorded and transcribed verbatim. The transcript were validated by re-listening to the tapes.

Constant comparative analysis was used for coding and category development. Incidents were identified in the data and coded. Initially, codes were identified as much as possible. Codes were compared to others codes. Codes were then collapsed into categories. In this process, incidents in a category were compared with previous incidents. New data was compared with data obtained earlier during the analysis phases. In intermediate coding, basic data was transformed into more abstract concepts allowing the theory to emerge from the data. Then, advanced coding was done to facilitate integration of the final grounded theory.

ELIGIBILITY:
Inclusion Criteria:

* care recipients having clinical diagnosis of dementia of any stage
* participants being the family caregivers of care recipients, providing care for at least 10 hours per week
* caregivers receiving case manager support for at least 3 months

Exclusion Criteria:

* caregivers who were under age of 18 and those exhibiting intellectual impairment
* caregivers who were not immediate family members of care recipients
* caregivers who could not communicate in Cantonese or English

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Family caregivers of person with dementia
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-05-02 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Semi-structured interview would be conducted individually | 2/5/2021-31/7/2021
  for data collection to explore the perspective of family caregivers on case manager approach in dementia care.

CONTACTS AND LOCATIONS:
Overall Officials: Kam Yan Lui, Miss, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Jockey Club Centre for Positive Ageing, Shatin, NT, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication. No identifying information about the individual would be revealed by using subject number
Supporting Information: Study Protocol, CSR
Time Frame: 3 years after completion and submission of study report
Access Criteria: Supporting information selected above will be shared to the public. Other supporting information will be accesible by principal investigator and academic supervisor only.